CLINICAL TRIAL: NCT03146923
Title: Decreasing Intakes & Absorption of Phosphorus in Haemodialysis Patients Through Food Choices
Acronym: DIP HD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Cork (Other)
Collaborators: Cork University Hospital (Other); Irish Nutrition & Dietetic Institute (Unknown)
Responsible Party: Principal Investigator, Joseph Eustace, Director of HRB Clinical Research Facility Cork, University College Cork
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17-CRFC-01
Record Dates: First submitted 2017-04-04; First posted 2017-05-10 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Renal Dialysis; Hyperphosphatemia; Dietary Modification
MeSH Terms: conditions — Hyperphosphatemia

STUDY DESIGN:
Intervention Model Description: Multicentre Parallel Arm Randomised Controlled Trial
Who Masked: Participant
Masking Description: As with most education based interventions compared to routine care it is difficult to reliably mask either the subjects or the investigators to the proposed intervention. We will attempt to blind patients referring only to the diets as diet A and diet B and avoiding the use of terminology such as old and new. We will reprint the dietary information for both arms so they do not resemble current illustrated formats.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care Arm (Active Comparator): Patients randomised to the standard care arm will be re educated using the current low phosphorus diet prescription.
  Interventions: Other: Current Low Phosphorus Diet Prescription
- Modified Intervention Arm (Experimental): Patients randomised to the intervention arm will be educated using a modified low phosphorus diet prescription.
  Interventions: Other: Modified Low Phosphorus Diet Prescription

INTERVENTIONS:
Other: Current Low Phosphorus Diet Prescription — Routine / Standard Care: Routine dietary intervention is currently provided by one-to-one counselling to the subject and his/her relevant family members or carers, by a state registered dietitian regarding a diet which provides <15mg Phosphorus /g Protein (over the day). This is equivalent to approximately 1000mg P / day. This is based on the 'Eating Well with Kidney Disease' dietsheet produced by the Renal Interest Group (RIG) of the Irish Nutrition & Dietetic Institute (INDI) in 2010 and includes following main components:
  * Restricting protein intake to requirements (1-1.2g/kg Ideal Body Weight)
  * Restricting dairy intake (1-1.5 portions per day)
  * Avoiding foods high in phosphate
  * Avoiding foods with phosphate additives
  Arms: Standard Care Arm
Other: Modified Low Phosphorus Diet Prescription — Modified Low Phosphorus Diet Prescription: The new prescription recommends five changes to current management
  * Introduction of some plant protein in the form of pulses and nuts where the phosphorus is largely bound by phytate
  * Increased focus on avoiding additives
  * Introduction of more whole grains e.g. wholemeal sliced pan/ pasta/rice .
  * Avoiding over-prescription of protein which carries an obligatory phosphorus load.
  * Focus on high protein foods with a low phosphorus to protein ratio
  Arms: Modified Intervention Arm

SUMMARY:
Based on new evidence renal dietitians in Ireland are revising the diet sheet that is used to teach patients about reducing blood phosphate. Changes that renal dietitians plan to make to the dietary phosphorus prescription

* Inclusion of some nuts and pulses
* More detailed education re phosphate additives
* More accurate protein prescription
* Inclusion of more whole grains
* Encouraging the use of foods with a low phosphorus to protein ratio

The investigators want to test the two diet prescription to find out, which one is better at reducing blood phosphate and which one is more acceptable to patients. The investigators also want to make sure it is safe.

DETAILED DESCRIPTION:
Background:

Chronic Kidney Disease (CKD) afflicts one in twenty Irish citizens who are over age 45 and is a significant risk factor for cardiovascular disease, premature death and significantly impacts healthcare utilisation. As kidney function deteriorates, phosphorus, upregulates counter regulatory hormones (immunoreactive Parathyroid Hormone (iPTH) and Fibroblast Growth Factor 23 (FGF23), the elevated levels of which are maladaptive. Collectively these abnormalities and their complications are referred to as Chronic Kidney Disease, Mineral & Bone Disorder (CKD MBD). Hyperphosphataemia or high blood phosphate levels is associated with increased mortality, in dialysis patients, in the earlier stages of CKD and even in patients with normal renal function. The use of phosphorus restricted diets in combination with oral phosphate binders has become well established in the management of patients with CKD stages 3-5 (including CKD stage 5D).

Experts have called for research into the dietary management of phosphate in the CKD population. The current evidence base is weak and in a recent Cochrane systematic review the authors concluded that there was limited low quality evidence to indicate that dietary interventions may positively affect CKD-MBD.

In recent years there has been increased focus on dietary phosphorus restriction in the management of CKD-MBD and a number of experts have suggested changes in how we manage dietary phosphorus. Several potential strategies have been suggested and in response the Renal Interest Group (RIG) of the Irish Nutrition & Dietetic Institute (INDI) held a 1 day meeting in Dublin in January 2015 which brought together numerous experts in the field to summarise our current understanding and the recent advances in the field.

Following on from this, RIG set up a working group to translate the new knowledge from the advanced study day and from further literature reviews into a modified low phosphate diet sheet.

Almost all people who have end stage kidney disease (ESKD) and require dialysis to survive, follow a dietary phosphorus restriction, to control high blood phosphate, with the aim of reducing the risk of cardiovascular disease, fractures and death.

Research Hypothesis: The modified low phosphate diet sheet is superior to current treatment in haemodialysis patients

Study Objectives

Primary Objective: To determine if the modified low phosphorus dietary prescription is superior to current management in reducing serum phosphate levels in HD patients

Secondary Objectives To determine if the modified low phosphorus diet is tolerable To determine if the modified low phosphorus diet is safe To determine if the modified low phosphorus diet brings the renal diet closer to healthy eating advice e.g. increased fibre intake.

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* Self reported urine output less than 2 cups (400mls) / day
* On maintenance haemodialysis for > 3 months
* Phosphate >1.6mmole/L on average of last 3 available routine monthly blood tests

Exclusion Criteria:

* Hyperkalemia, defined as a predialysis serum K on routine monthly blood test of >6mmoles/l in the month preceding the trial.
* Parathyroidectomy
* Corrected serum calcium <2.2 or > 2.6mmol/L or local normal units where ranges varied significantly from 2.2-2.6mmoles/l.
* Acute concurrent illness, requiring hospitalisation in the 2 weeks prior to recruitment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2017-06-16 (Actual); Study Completion 2017-06-16 (Actual)

PRIMARY OUTCOMES:
Serum Phosphate | 1 month
  Difference in serum phosphate value at 1 month v baseline, in those randomised to the modified diet compared to the difference in serum phosphate value at 1 month v baseline in those randomised to standard care.

SECONDARY OUTCOMES:
Dietary Intake | 1 month
  Between arm difference in dietary phosphate intake (separating phosphate into high & low bioavailability).
  Between arm difference in dietary fibre intake.
Serum iPTH | 1 month
  Difference in serum iPTH value at 1 month v baseline, in those randomised to the modified diet compared to the difference in serum iPTH value at 1 month v baseline in those randomised to standard care.
Palatability and Subject Acceptance (Tolerability) | 1 month
  Palatability and subject acceptance of modified diet as assessed by 5 point Likert Scale
FGF23 (Exploratory Endpoint) | 1 month
  Within subject change in geometric mean FGF-23 measurement at baseline as compared to the end of the 1 month intervention. Because of evidence that subjects with diabetes handle phosphorus differently we will analyse result for FGF 23 separately in patients with and without diabetes (Muras et al., 2013, Yoda et al., 2012).
Serum Potassium (Safety Endpoints): | 1 month
  Check serum potassium in week 2. Difference in serum potassium value at 1 month v baseline, in those randomised to the modified diet compared to the difference in serum potassium value at 1 month v baseline in those randomised to standard care.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Eustace, MB, Principal Investigator — HRB Clinical Research Facility
Locations (10):
- Ireland (10):
  - Midland Regional Hospital Tullamore, Tullamore, Offaly
  - Cavan General Hospital, Cavan
  - Fiona Byrne, Cork
  - St. Vincents University Hospital, Dublin
  - Mater Misericordia University Hospital, Dublin
  - Beaumont Hospital, Dublin
  - Tallaght Hospital, Dublin
  - Galway University Hospitals, Galway
  - University Hospital Limerick, Limerick
  - Mayo University Hospital, Mayo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Byrne F, Gillman B, Renal Interest Group INDI, Eustace J. Multicentre Randomized Control Trial of Phosphate Control with a Modified as Compared to Standard Renal Diet TH-OR030. J Am Soc Nephrol 2018;29:8.
- See also: Link to abstract of oral presentation at the American Society of Nephrology's 2018 Kidney Week — https://www.asn-online.org/education/kidneyweek/2018/program-abstract.aspx?controlId=3024392